CLINICAL TRIAL: NCT06681324
Title: A Participant- and Investigator-blind, Randomized, Placebo-controlled Phase II Study to Evaluate Safety, Tolerability, and Mucosal Repair With AZD7798 in Patients With Active Ileal Crohn's Disease and an Ileostomy (CALLISTO)
Brief Title: Study Evaluating AZD7798 for Treatment in Crohn's Disease Patients With an Ileostomy
Acronym: CALLISTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: D9690C00006
Record Dates: First submitted 2024-09-25; First posted 2024-11-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; ileostomy; inflammation; small bowel; stoma
MeSH Terms: conditions — Crohn Disease; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to receive either AZD7798 or placebo during 12-week participant- and Investigator- blind induction period. At week 12 after induction period, all eligible participants will enter 40-week open label maintenance period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD7798 (Experimental): AZD7798
  Interventions: Drug: AZD7798
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD7798 — AZD7798
  Arms: AZD7798
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, and effect on mucosal repair of AZD7798 compared with placebo in participants with active ileal Crohn's disease and an ileostomy.

DETAILED DESCRIPTION:
This is a participant-and investigator-blind, randomized, parallel-group, placebo controlled phase II study designed to evaluate safety, tolerability, and mucosal repair with AZD7798 in participants with active ileal Crohn's disease and an ileostomy. This study will include a screening period, an induction period, an open-label maintenance period, and a follow-up period. Approximately 30 participants will be randomized globally to receive either AZD7798 or placebo during 12-week participant- and investigator- blind induction period. At week 12 after induction period, all eligible participants will enter 40-week open label maintenance period. Follow-up visits will take place 8 weeks and 18 weeks after the last dose of study intervention, whether this occurs during the induction period or the open-label maintenance period.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age.
* Diagnosis of Crohn's disease established with clinical, imaging, endoscopic, and/or histopathologic evidence.
* Ileostomy for at least 3 months.
* Prior to screening endoscopy, clinical suspicion of active ileal inflammation based on at least one of the following: previous endoscopy, imaging (CT, MRI, IUS), or FCP above upper reference limit.
* Active ileal Crohn's disease as determined by active intestinal mucosal inflammation, as demonstrated on video recorded ileoscopy performed during the screening period and scored by a blinded central reader with agreement on the SES CD ≥ 4 of the ileal segment proximal to the stoma. Participants with inflammation in additional intestinal segments are not excluded.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Concomitant additional gastrointestinal luminal inflammatory diseases
* Strictures/stenoses preventing passage of endoscope throughout the specified segment
* Short bowel syndrome
* Within 3 months prior to screening:

  1. Diagnosis of peritonitis or need treatment of peritonitis
  2. Bowel perforation or evidence of obstruction
* All intrabdominal, cutaneous and perianal/perirectal abscesses and fistulae are excluded with exception of: cutaneous and perianal/perirectal abscesses which are adequately drained 4 weeks prior to randomization, and intraabdominal fistulae between bowel segments only without complications
* Ongoing or expected nutritional dependency on total enteral or parenteral nutrition during study (partial nutrition acceptable).
* In participants with any remaining colon and/or rectum, evidence of an increased risk of colorectal cancer, including:

  1. Adenomatous colonic/rectal polyps that have not been removed
  2. Intestinal dysplasia
  3. Not undertaking appropriate surveillance, if indicated, for colorectal dysplasia/malignancy
* Reversal of ileostomy or formation of J-pouch planned prior to end of study period.
* High-output stoma (eg, > 2000 mL/24 hours) associated with volume depletion and/or electrolyte disturbance to the extent that, in the opinion of the Investigator, it may put the participant at undue risk because of participation in the study, or impact their ability to participate in the study or interfere with the interpretation of study data.
* Any of the following treatments within the specified time period:

  1. An anti-TNF biologic within 8 weeks prior to randomization
  2. Any biologic targeting immune response other than an anti-TNF (including vedolizumab and ustekinumab) within 12 weeks prior to randomization.
  3. Other advanced small molecule treatments for Crohn's disease within 4 weeks prior to randomization
  4. Cyclosporine, mycophenolate mofetil, sirolimus (rapamycin), thalidomide, or tacrolimus within 4 weeks prior to randomization
  5. Treatment with apheresis (eg, Adacolumn, Cellsorba) within 4 weeks prior to randomization
  6. Administration of any live vaccine within 4 weeks prior to randomization, or planned administration of any such vaccine during the study
  7. Faecal microbiota transplantation within 4 weeks prior to randomization
  8. Regular intake of NSAIDs within 12 weeks prior to screening ileoscopy and during the study (defined as at least times per week for more than 3 months; not applicable to daily aspirin use up to 325 mg per day)
  9. Lymphocyte-depleting treatment, including, but not limited to rituximab, within 12 months prior to randomization
* Any changes in dosing of the following medications prior to screening ileoscopy as outlined

  1. 5-aminosalicylates within 2 weeks
  2. Oral corticosteroids within 2 weeks. Also excluded if on stable dosing of steroids exceeding the following dose equivalents:

  (i) Systemic steroids > 20 mg/day prednisolone dose or equivalent (ii) Locally targeted steroids exceeding maximum budesonide dose or equivalent [9 mg/day] (c) Immunomodulators (thiopurines or methotrexate) within 4 weeks (d) Antibiotic therapy for the treatment of Crohn's disease, eg, ciprofloxacin or metronidazole within 2 weeks (e) Probiotics within 2 weeks
* Evidence of recent or currently active infection, including use of IV or oral antibiotics for documented infection within 30 days prior to screening.
* Evidence of chronic hepatitis B or C infection
* History of TB (active or latent) unless an appropriate course of treatment has been completed.
* Positive diagnostic TB test at screening.
* History of serious opportunistic infection within 12 months prior to screening
* Symptomatic herpes zoster infection within 3 months prior to screening.
* Positive C. difficile toxin test at screening.
* Any identified immunodeficiency
* Any other abnormal laboratory results at screening, which, in the opinion of the Investigator, will prevent the participant from completing the study or will interfere with the interpretation of the study results
* Prolonged QTcF interval > 450 ms (or > 480 ms for patients with bundle branch block) or congenital long-QT syndrome or family history of long-QT syndrome or sudden cardiac death in age < 40 years.
* Clinically significant cardiovascular conditions
* Reproduction:

  1. Pregnant and breastfeeding participants, or those planning to breastfeed during the study
  2. FOCBP, unless they agree to complete abstinence or to use a highly effective contraceptive method AND barrier method
* Current malignancy or history of malignancy
* Current significant major or unstable respiratory disease, heart disease, cerebrovascular disease, haematological disease, hepatic disease including large duct primary sclerosing cholangitis with jaundice, recurrent cholangitis or cirrhosis, renal disease, gastrointestinal disease, or other major disease other than active Crohn's disease.
* Current enrolment in another interventional study or treatment with any investigational drug within 4 months (or 5 half-lives, whichever is longer) prior to screening
* Unstable lifestyle factors
* Participants committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
* Involvement in the planning and/or conduct of the study
* Judgement by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
* Previous randomization in the present study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2027-06-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | from Week 0 to Week 12
  Summary of any adverse events and also by MedDRA SOC and Preferred term
Number of participants with abnormal Vital signs: Blood pressure | from Week 0 to Week 12
  Systolic and diastolic blood pressure will be summarized by descriptive statistics
Number of participants with abnormal Vital signs: Pulse rate | from Week 0 to Week 12
  Pulse rate will be summarized by descriptive statistics
Number of participants with abnormal values in haematology: complete blood count (CBC) | from Week 0 to Week 12
  The variables platelet count, red blood cell (RBC) count, haemoglobin, haematocrit will be summarized with descriptive statistics
Number of participants with abnormal values in haematology: white blood cell (WBC) count | from Week 0 to Week 12
  The variables neutrophils, lymphocytes, monocytes, eosinophils, and basophils will be summarized with descriptive statistics
Number of participants with abnormal values in haematology: RBC | from Week 0 to Week 12
  The variables mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH) and percentage of reticulocytes will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: kidney function | from Week 0 to Week 12
  The variables creatinine and blood urea nitrogen (BUN) will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: electrolytes | from Week 0 to Week 12
  The variables potassium, sodium, and calcium will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: liver function | from Week 0 to Week 12
  The variables ALT (Alanine Aminotransferase), AST (Aspartate Aminotransferase), and ALP (alkaline phosphatase), and albumin will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: hs-CRP | from Week 0 to Week 12
  The variable hs-C-reactive protein will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: glucose | from Week 0 to Week 12
  The variable glucose will be summarized with descriptive statistics
Number of participants with abnormal values in ECG readings | from Week 0 to Week 12
  12-lead ECGs will be obtained using an ECG machine, that automatically measures RR/HR, PR, QRS, QT and Corrected QT (QTc) intervals, and summarized with descriptive statistics

SECONDARY OUTCOMES:
Difference in mean change from baseline in endoscopic score between active and placebo | Week 12
  Simple Endoscopic Score for Crohn's Disease (SES-CD) is based on the evaluation of ileum, and the presence and size of ulcerations and the extent of the inflammatory area and stenosis are assessed. The segment is scored from 0 to 12, higher scores indicating more active disease
Number of participants with endoscopic response | Week 12
  Endoscopic response is defined as ≥ 50% decrease from baseline in SES-CD total score and based on the evaluation of ileum and the presence and size of ulcerations and the extent of the inflammatory area and stenosis are assessed. The segment is scored from 0 to 12, higher scores indicating more active disease
Number of participants with endoscopic remission | Week 12
  Endoscopic remission is defined as SES-CD total score < 4 and at least 2 point reduction from baseline with no sub score > 1 in any individual variable. SES-CD is based on the evaluation of ileum, and the presence and size of ulcerations and the extent of the inflammatory area and stenosis are assessed. The segment is scored from 0 to 12, higher scores indicating more active disease
Serum AZD7798 concentration | up to 52 Weeks
  Serum AZD7798 concentration (PK)
Incidence of anti-drug antibody response | up to 52 Weeks
  Incidence of anti-drug antibody (ADA) response - number and percentages with a positive ADA result
Titre of anti-drug antibody response | up to 52 Weeks
  Titre of anti-drug antibody (ADA) response - immunogenicity titre will be summarized descriptively as a continuous variable, only for ADA positive tests
Number of participants with adverse events in active treatment | from Week 12 to Week 52
  Summary of any adverse events and also by MedDRA SOC and Preferred term
Number of participants with abnormal vital signs: Blood pressure | from Week 12 to Week 52
  Systolic and diastolic blood pressure will be summarized by descriptive statistics
Number of participants with abnormal vital signs: Pulse rate | from Week 12 to Week 52
  Pulse rate will be summarized by descriptive statistics
Number of participants with abnormal values in haematology: complete blood count (CBC) | from Week 12 to Week 52
  The variables platelet count, red blood cell (RBC) count, haemoglobin, haematocrit will be summarized with descriptive statistics
Number of participants with abnormal values in haematology: white blood cell (WBC) count | from Week 12 to Week 52
  The variables neutrophils, lymphocytes, monocytes, eosinophils, and basophils will be summarized with descriptive statistics
Number of participants with abnormal values in haematology: RBC | from Week 12 to Week 52
  The variables mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH) and percentage of reticulocytes will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: kidney function | from week 12 to week 52
  The variables creatinine and blood urea nitrogen (BUN) will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: electrolytes | from Week 12 to Week 52
  The variables potassium, sodium, and calcium will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: liver function | from Week 12 to Week 52
  The variables ALT (Alanine Aminotransferase), AST (Aspartate Aminotransferase), and ALP (alkaline phosphatase), and albumin will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: hs-CRP | from Week 12 to Week 52
  The variable hs-C-reactive protein will be summarized with descriptive statistics
Number of participants with abnormal values in clinical chemistry: glucose | from Week 12 to Week 52
  The variable glucose will be summarized with descriptive statistics
Number of participants with abnormal values in ECG readings | from week 12 to week 52
  12-lead ECGs will be obtained using an ECG machine, that automatically measures RR/HR, PR, QRS, QT and Corrected QT (QTc) intervals, and summarized with descriptive statistics

CONTACTS AND LOCATIONS:
Locations (18):
- Research Site, Leuven, Belgium
- Italy (3):
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
- Poland (4):
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Stockholm
- Ukraine (2):
  - Research Site, Kyiv
  - Research Site, Vinnytsia
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/